CLINICAL TRIAL: NCT01114828
Title: A Multi-center, Double-blind, Parallel-arm Study to Investigate Pharmacodynamics and Pharmacokinetics of OPC-41061 in Patients With Hepatic Edema
Brief Title: A Study to Investigate Pharmacodynamics and Pharmacokinetics of OPC-41061 in Patients With Hepatic Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-09-004; JapicCTI-101112 (Other: JAPIC)
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; ascites; Tolvaptan; OPC-41061
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3.75 mg (Experimental): Once-daily oral administration of OPC-41061
  Interventions: Drug: OPC-41061
- 7.5 mg (Experimental): Once-daily oral administration of OPC-41061
  Interventions: Drug: OPC-41061

INTERVENTIONS:
Drug: OPC-41061 — Once-daily oral administration of OPC-41061 at 3.75 mg after breakfast for 7 days
  Arms: 3.75 mg
Drug: OPC-41061 — Once-daily oral administration of OPC-41061 at 7.5 mg after breakfast for 7 days
  Arms: 7.5 mg

SUMMARY:
OPC-41061 at 3.75 mg/day or 7.5 mg/day will be orally administered once daily for 7 days to cirrhosis patients with ascites despite having received treatment with conventional diuretics and pharmacodynamics, pharmacokinetics, efficacy, and safety will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients judged as having cirrhosis based on previous imaging diagnosis (Definition of cirrhosis includes patients with collateral circulation due to chronic hepatic impairment)
* Patients with ascites in whom the dose of existing diuretics cannot be increased due to risk of adverse drug reactions such as electrolyte abnormalities, or in whom sufficient therapeutic effect cannot be obtained with existing diuretics
* Patients who have been receiving oral combination therapy with a loop diuretic and an anti-aldosterone agent from at least 7 days prior to receipt of informed consent, with a dose combination of either loop diuretic equivalent to furosemide 40 mg/day or higher plus spironolactone 25 mg/day or higher, or loop diuretic equivalent to furosemide 20 mg/day or higher plus spironolactone 50 mg/day or higher
* Patients who are hospitalized or who can be hospitalized for the trial - Age 20 to 80 years inclusive
* Patients capable of giving informed consent
* Patients who, together with their partner, agree to use an appropriate method of contraception until 4 weeks after the final trial drug administration

Exclusion Criteria:

* Patients with any of the following complications or symptoms:

  * Hepatic encephalopathy (hepatic coma of grade 2 or higher)
  * Hepatocellular carcinoma with imaging-diagnosed vascular infiltration into trunk or primary branch of portal vein, inferior vena cava, or trunk of hepatic vein
  * Endoscopic findings from screening examination or from within 30 days prior to screening examination indicating the need for new therapy for esophageal or gastric varices during the trial period
  * Repeated hemorrhoidal bleeding due to rectal varicose veins within 30 days prior to informed consent
  * Heart failure (New York Heart Association Class III or IV)
  * Anuria
  * Impaired urination due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
* Patients with a history of any of the following disorders:

  * Cerebrovascular disorder within 30 days prior to informed consent
  * Hypersensitivity or idiosyncratic reaction to benzazepine derivatives (such as mozavaptan hydrochloride or benazepril hydrochloride) "
* Morbidly obese patients with a body mass index (BMI: body weight (kg)/height (m)2) exceeding 35
* Patients with sitting systolic blood pressure lower than 90 mm Hg
* Patients with any of following abnormal clinical laboratory values at time of the screening examination: Hemoglobin lower than 8.0 g/dL, total bilirubin higher than 4.0 mg/dL, serum creatinine higher than 2.0 mg/dL, serum sodium higher than 147 mEq/L, or serum potassium higher than 5.5 mEq/L
* Patients who are unable to take oral medication
* Female patients who are pregnant, possibly pregnant, or breast-feeding, or who are planning to become pregnant
* Patients who have used albumin preparations (therapeutic agents for hypoalbuminemia) or blood products containing albumin from within 7 days prior to informed consent
* Patients who received any investigational drug other than OPC-41061 within 30 days prior to informed consent
* Patients who have previously received OPC-41061
* Any patient who, in the opinion of the principle investigator or subinvestigator, is inappropriate for participation in the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Department of Clinical Research and Development, Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Tokyo, Et Al., Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- 3.75 mg: Once-daily oral administration of OPC-41061 at 3.75 mg after breakfast for 7 days
- 7.5 mg: Once-daily oral administration of OPC-41061 at 7.5 mg after breakfast for 7 days
Period: Overall Study
Arm/Group | 3.75 mg | 7.5 mg
Started | 19 | 21
Completed | 16 | 17
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.75 mg | 7.5 mg | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.3) | 64.2 (10.4) | 65.7 (9.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 11 | 18
  >=65 years | 12 | 10 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  Japan | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Changes from baseline (day-1) for body weight at the end of treatment (LOCF) were calculated.
Time Frame: Bseline, Day 7 or at the discontined of treatment
Population: For efficacy analysis set, 3 participants of 3.75 mg arm were excluded by violation of protocol and one participant of 7.5 mg arm was excluded by concomitant edematous disorders other than hepatic.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- OPC-41061 3.75 mg: Once-daily oral administration of OPC-41061 at 3.75 mg after breakfast for 7 days
- OPC-41061 7.5 mg: Once-daily oral administration of OPC-41061 at 7.5 mg after breakfast for 7 days
Arm/Group | OPC-41061 3.75 mg | OPC-41061 7.5 mg
Number analyzed (Participants) | 16 | 20
kg | -1.14 (0.86) | -1.37 (2.05)

2. Secondary Outcome: Ascites Volume as Measured by CT
Description: Change from baseline (day-1) for ascites volume as measured by CT at the end of treatment (LOCF) were calculated.
Time Frame: Baseline, Day 7 or at the discontinued of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | OPC-41061 3.75 mg | OPC-41061 7.5 mg
Number analyzed (Participants) | 16 | 20
mL | -407.5 (545.8) | -514.0 (993.8)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | 3.75 mg | 7.5 mg
Serious Adverse Events (participants affected / at risk) | 2/19 | 3/21
Other Adverse Events (participants affected / at risk) | 13/19 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75 mg (N=19) | 7.5 mg (N=21)
Gastrointestinal Angiodysplasia Haemorrhagic (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood Potassium Increased (Investigations) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75 mg (N=19) | 7.5 mg (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (1)
Reflux Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (2)
Thirst (General disorders) | 3 (3) | 7 (7)
Pylethrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Colitis Pseudomembranous (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (2) | 0 (0)
Blood Glucose Decreased (Investigations) | 0 (0) | 1 (1)
Blood Potassium Increased (Investigations) | 2 (3) | 0 (0)
Blood Pressure Decreased (Investigations) | 3 (4) | 0 (0)
Blood Sodium Decreased (Investigations) | 1 (1) | 0 (0)
Blood Urea Increased (Investigations) | 0 (0) | 1 (1)
Blood Urine Present (Investigations) | 2 (2) | 1 (1)
Prothrombin Time Prolonged (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No